CLINICAL TRIAL: NCT01789385
Title: Anesthesia for Deep Brain Stimulation for the Treatment of Parkinsons Disease
Brief Title: Anesthesia for Deep Brain Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, MD, Diskapi Teaching and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DİLEKPARKİNSON
Record Dates: First submitted 2013-02-02; First posted 2013-02-12 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2013-02

CONDITIONS: Parkinsons Disease
Keywords: Deep brain stimulation; Parkinson
MeSH Terms: conditions — Parkinson Disease | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dexmedetomidine (Other): Precedex 200 mcg 2ml
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Starting with a 1 mg kg-1min-1 loading dose and than continued with a0.2-0.8 mg kg-1h-1 infusion rate.
  Other Names: Precedex 200 mcg 2 ml

SUMMARY:
Deep brain stimulation for the treatment of Parkinson's disease has unique surgical stages and anesthesia needs. In the first stage the electrodes are inserted in the targeted brain areas and in the second stage the pulse generator is implanted. The technique for establishing sedation and analgesia for functional neurosurgery may differ among institutions. In this study it was aimed to investigate our anesthesia methods, intra-operative adverse events in the first stage of deep brain stimulation and the post operative pain therapy of the patients.

DETAILED DESCRIPTION:
This study included patients underwent deep brain stimulation (DBS) in the treatment of patients with Parkinson disease (PD). After obtaining ethical approval and patient consent, consecutive patients underwent deep brain stimulation with a predetermined anesthesia protocol were studied.

The anesthetic procedure was explained to the patients in detail by the responsible anesthetist. Patients requiring general anesthesia, suffering from dementia, obstructive sleep apnea, gastroesophageal reflux and with a mallampati score>2, musculoskeletal problems causing difficulty with long term surgical positioning were excluded. The following parameters were recorded:Gender, age, body mass index (BMI), ASA classification, co existing diseases, anti Parkinson medications, sedative drugs and doses, level of conscious sedation, local anesthetic agents and doses, total duration of procedure, adverse events and complications, post operative pain therapy.

Preoperative sedation was not administered. At arrival in the operating room patients were monitored for heart rate (HR) non invasive blood pressures (systolic arterial pressure; SAP, diastolic arterial pressure; DAP, mean arterial pressure; MAP) peripheral oxygen saturation (SPO2), respiratory rate (RR), BIS, baseline values were recorded and recordings were continued with 5 min intervals. Urinary catheterization was not applied. Adequate attention was payed to assure all patients to be in a comfortable position. A peripheral intravenous catheter was inserted and Ringers lactate solution was infused 50-100 ml h-1. All patients received oxygen 2 L min-1 via a nasal cannula. Nasal airway, LMA and ET was prepared as rescue airway devices. Periods of SPO2 < 92 and a RR ≤ 8 min were documented. Maneuvers needed to manipulate airway patency was recorded. A 20% difference in the initial hemodynamic parameters and the use of hypotensive or inotrope, vasopressor medications were recorded.

Initial sedation was employed with a 1 mg kg-1min-1 loading dose of dexmedetomidine (Precedex®,Hospira Inc, Rocky Mountain, USA) for 10 minutes. Sedation was maintained with dexmedetomidine at a 0.2-0.8 mg kg-1h-1 infusion rate. Invasive blood pressure monitoring will be applied after sedation is commenced. After achieving an adequate sedation level which is defined as a BIS value of 65-85 and the Ramsay sedation score 3, the scalp block was performed as previously described by Girvin. A superficial cervical plexus block was also performed. Bupivacaine was used for the nerve blocks. Lidocaine was used for local anesthetic scalp infiltration in case of insufficient analgesia was observed during the insertion of the head pins or at any time the patient complained having pain. Ephedrine 1/200000 was added to the local anesthetics. Local anesthetic agents were diluted with equivalent volumes of saline (1/1 volume). The total doses of local anesthetics was recorded at the end of the procedure. Propofol was used with incremental intravenous boluses for rescue sedation when needed and the total dose will be documented. Sedation was discontinued before the micro electrode recordings (MER's) and macro stimulation. Time to emergence was defined as the time between the discontinuation of the sedatives and the time between the patients are able to cooperate with the neurologic examination. All intra-operative events and complications and complaints regarding pain and restlessness were documented. The total duration of the procedure includes initial sedation, performance of regional anesthesia, stereotactic frame insertion, magnetic resonance (MRI) or computerized tomography (CT) imaging, MER's, macro stimulation and closure.

After completion of procedure patients were transferred to the post anesthesia care unit (PACU). Postoperative pain was evaluated in the PACU at arrival and then at 1, 6, 12, 24 h using a 0-10 cm verbal analog scale (VAS)(zero: no pain, 10: maximal pain). Patients received 50 mg tramadol 8 hourly and PCA with morphine(5 mg loading dose, 2 mg bolus, 15 min lockout time) was initiated when the VAS ≥ 3. Morphine consumption was measured at 24 h.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing DBS for the treatment of PD

Exclusion Criteria:

* Patients required general anesthesia,
* suffered from dementia,
* obstructive sleep apnea,
* gastro esophageal reflux and with a mallampati score > 2,
* musculoskeletal problems causing difficulty with long term surgical positioning were excluded.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Doses of the sedative agents | 1 day
  Dexmedetomidine, propofol and midazolam will be used for sedation. We will determine the doses needed to tolerate surgery and to allow MER's and macrostimulation

SECONDARY OUTCOMES:
Time to emergence | 1 day
  time from discontinuation of sedative drugs to time that the patients are able to cooperate with macrostimulation

OTHER OUTCOMES:
postoperative pain scores | postopertive 1 day
  visual analog pain scores of the patients at postoperative 1, 6, 12 and 24th hours

CONTACTS AND LOCATIONS:
Overall Officials: Dilek YAZICIOGLU, MD, Principal Investigator — Ankara Diskapi Yildirim Beyazit Teaching and Research Hospital, Turkey.
Locations (1):
- Ankara Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Genty S, Derrey S, Pouplin S, Lefaucheur R, Chastan N, Gerardin E, Maltete D. Pain due to osteoarthritis may impair the early outcome of deep brain stimulation in Parkinson's disease. Clin Neurol Neurosurg. 2011 Dec;113(10):864-7. doi: 10.1016/j.clineuro.2011.06.006. Epub 2011 Jul 19. PMID 21775052
- [Background] Yagar S, Yavas S, Karahalil B. The role of the ADRA2A C1291G genetic polymorphism in response to dexmedetomidine on patients undergoing coronary artery surgery. Mol Biol Rep. 2011 Jun;38(5):3383-9. doi: 10.1007/s11033-010-0446-y. Epub 2010 Nov 23. PMID 21104443
- [Result] Stoneham MD, Cooper R, Quiney NF, Walters FJ. Pain following craniotomy: a preliminary study comparing PCA morphine with intramuscular codeine phosphate. Anaesthesia. 1996 Dec;51(12):1176-8. doi: 10.1111/j.1365-2044.1996.tb15065.x. PMID 9038464